CLINICAL TRIAL: NCT01535040
Title: Randomized Placebo-Controlled Phase 2 Pilot Study of Memantine (Namenda) for Smoking Cessation Among Cancer Survivors
Brief Title: Memantine Hydrochloride in Helping Cancer Survivors Stop Smoking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRB00020412; U10CA081851 (NIH); REBACCCWFU 99311 (Other: NCI)
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Prostate Cancer; Tobacco Use Disorder
Keywords: cancer survivor; stage I non-small cell lung cancer; stage II non-small cell lung cancer; tobacco use disorder; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage I prostate cancer; stage IIA prostate cancer; stage IIB prostate cancer; stage III prostate cancer; stage I colon cancer; stage IIA colon cancer; stage IIB colon cancer; stage IIC colon cancer; stage IIIA colon cancer; stage IIIB colon cancer; stage IIIC colon cancer; stage I rectal cancer; stage IIA rectal cancer; stage IIB rectal cancer; stage IIC rectal cancer; stage IIIA rectal cancer; stage IIIB rectal cancer; stage IIIC rectal cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Tobacco Use Disorder; Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Rectal Neoplasms | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I - Memantine (Active Comparator): Participants receive memantine hydrochloride PO BID) on days 1-81 in the absence of unacceptable toxicity.
  Interventions: Drug: memantine hydrochloride
- Arm II - Placebo (Placebo Comparator): Participants receive a placebo PO BID on days 1-81 in the absence of unacceptable toxicity.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: memantine hydrochloride — Estimate participation, accrual, adherence, and retention of cancer survivors who smoke and are randomized to receive memantine (10 mg twice daily) or a matching placebo for 12 weeks.
  Other Names: Memantine
  Arms: Arm I - Memantine
Drug: placebo — Placebo by mouth through completion of 12 weeks.
  Arms: Arm II - Placebo

SUMMARY:
RATIONALE: Memantine hydrochloride may help people stop smoking by decreasing the symptoms of nicotine withdrawal.

PURPOSE: This randomized, pilot phase II trial studies how effective memantine hydrochloride works compared to placebo in helping cancer survivors stop smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate participation, accrual, adherence, and retention of cancer survivors who smoke and are randomized to receive memantine (memantine hydrochloride) (10 mg twice daily) or a matching placebo for 12 weeks.
* Estimate the self-reported abstinence rates of patients who are randomized to memantine or a matching placebo for 12 weeks and obtain a preliminary estimate of the treatment effect (difference in abstinence rates between the two groups).

Secondary

* Nicotine addiction will be assessed using the Wisconsin Inventory of Smoking Dependent Motives.
* Nicotine withdrawal will be measured by the Wisconsin Smoking Withdrawal Scale.
* Quality of life will be measured by the SF12 questionnaire.
* Toxicities will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.

OUTLINE: This is a randomized, placebo-controlled, pilot study. Participants are stratified according to gender (male vs female). Participants are randomized to 1 of 2 treatment arms.

* Arm I: Participants receive memantine hydrochloride orally (PO) twice daily (BID) on days 1-81 in the absence of unacceptable toxicity.
* Arm II: Participants receive placebo PO BID on days 1-81 in the absence of unacceptable toxicity.

Participants complete the Behavioral Risk Factor Surveillance Survey (BRFSS), the Self-reported Tobacco Abstinence, the Wisconsin Inventory of Smoking Dependent Motives, the Wisconsin Smoking Withdrawal Scale, SF-12 quality-of-life questionnaire, and the Fagerstrom Nicotine Tolerance Scale at baseline and every 2 weeks for 12 weeks during study.

Participants also undergo urine sample collection at weeks 4, 8, and 12 for cotinine test using the NicAlert test.

ELIGIBILITY:
INCLUSION CRITERIA:

* Survivors of non-metastatic breast, prostate, or colorectal cancer, or stage I/II non-small cell lung cancer
* Age ≥ 18
* Smoked 100 tobacco cigarettes over lifetime at time of first interview, have smoked 10 or more cigarettes per day on most days over the past month
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky ≥ 70%)
* Ability to understand and the willingness to sign a written informed consent document
* Agrees to adhere to the study protocol and attend the required clinic visits
* Negative serum pregnancy test within 10 days prior to registration in women with child-bearing potential; women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Women who are currently breast-feeding are not eligible for this study

Exclusion Criteria:

* Use of chewing tobacco, pipe tobacco, snuff, or any other non-cigarette tobacco product is not allowed
* No patients with clinically significant uncontrolled medical conditions (e.g., unstable angina, myocardial infarction, transient ischemic attack [TIA], or cerebral vascular accident [CVA]) within past 3 months
* Creatinine ≥ 2 times upper limit of normal (ULN) in last six months
* Serum glutamic oxaloacetic transaminase (SGOT)/serum glutamic pyruvate transaminase (SGPT) ≥ 3 times ULN in last six months
* Current uncontrolled hypertension ≥ 160/90 mm Hg
* Excessive alcohol abuse defined as more than 5 drinks per day for men and 4 drinks per day for women
* Major medical or psychiatric illness which, in the opinion of the investigator, would prevent completion of treatment or would interfere with follow-up
* History of allergic reactions attributed to memantine

PRIOR CONCURRENT THERAPY:

* Six months post definitive treatment (except for ongoing hormonal or targeted therapies)
* Patients currently must not be taking Nicotine Replacement Therapy (NRT) and agree to not start NRT for the duration of the study
* Patients currently taking antidepressant or antianxiety medications must have been on a stable dose for 4 weeks prior to registration
* Patients currently receiving the following medications are not eligible: anticonvulsant agents (e.g., phenytoin, carbamazepine, gabapentin, etc.); antiparkinsonian agents (e.g., Levo Dopa, ropinirole); neuroleptic agents (e.g., risperidone, quetiapine); carbonic anhydrase inhibitors (e.g., Diamox® and Sequels®)
* Memantine should not be combined with other N-methyl d-aspartate (NMDA) antagonists (amantadine, ketamine, and dextromethorphan)
* Participants may not be receiving any other investigational agents
* No current use of illegal drugs or use of prescription medications for non-medical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2014-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Spangler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Cancer Center CCOP Research Base, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Spangler J, Skidmore E, Dressler EV, Weaver KE, Lesser GJ, Burton G, Esparaz B, Gillett B, Shaw EG. Randomized Placebo-Controlled Trial of Memantine for Smoking Cessation (CCCWFU 99311). Cancer Control. 2025 Jan-Dec;32:10732748251336416. doi: 10.1177/10732748251336416. Epub 2025 May 8. PMID 40340434

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I - Memantine | Arm II - Placebo
Started | 65 | 65
Completed | 35 | 44
Not Completed | 30 | 21
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 13 | 10
Not completed — Never Started | 9 | 4
Not completed — Toxicity | 7 | 5
Not completed — Multiple Reasons | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Memantine | Arm II - Placebo | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 54 | 100
  >=65 years | 19 | 11 | 30
Age, Continuous [Median (Full Range); unit: years] | 57 [29 to 84] | 56 [31 to 76] | 57 [29 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 110
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 65 | 64 | 129
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 11 | 18
  White | 58 | 53 | 111
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 65 | 65 | 130

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Retention is defined as the percentage of participants who complete the 12 week visit
Time Frame: 12 weeks
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I - Memantine | Arm II - Placebo
Number analyzed (Participants) | 65 | 65
percentage of participants | 53.8 [41.0 to 66.3] | 67.7 [54.9 to 78.8]

2. Primary Outcome: Adherence
Description: Adherence is the percentage of prescribed pills taken while on therapy.
Time Frame: 12 weeks
Population: Participants who returned pill diaries.
Measure: Mean (Full Range); unit: percentage of prescribed pills
Arm/Group | Arm I - Memantine | Arm II - Placebo
Number analyzed (Participants) | 48 | 52
percentage of prescribed pills | 86.0 [0 to 100] | 93.0 [10 to 100]

3. Secondary Outcome: Nicotine Dependence
Description: The Fagerstrom tolerance scale consists of 8 questions, each of which is scored on a 0 to 1 or 0 to 2 scale. The total score ranges from 0 to 11, with higher scores representing greater dependence.
Time Frame: 12 weeks
Population: Participants who reported any data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I - Memantine | Arm II - Placebo
Number analyzed (Participants) | 64 | 65
units on a scale | 5.29 (0.30) | 4.83 (0.28)

4. Secondary Outcome: Smoking Withdrawal
Description: The Wisconsin Smoking Withdrawal Scale is a 28 item questionnaire that assesses nicotine withdrawal. It consists of seven subscales, each consisting of 3-5 questions all answered on a 0-4 scale. Subscale scores are the mean of the items comprising the scale. Some items are reverse scored. Higher scores indicate greater withdrawal symptoms. Subscales were scored if more than half the items were answered. A total score was calculated as the mean of the individual subscales (if more than half the subscales had scores).
Time Frame: 12 weeks
Population: Participants who provided data at any time
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I - Memantine | Arm II - Placebo
Number analyzed (Participants) | 63 | 64
units on a scale | 1.93 (0.09) | 2.01 (0.08)

ADVERSE EVENTS:
Time Frame: 4 months (3 months of treatment and 1 month following the end of treatment)
Description: The sample size for this section is the number of participants who had post-randomization toxicity data recorded.
Arm/Group | Arm I - Memantine | Arm II - Placebo
Serious Adverse Events (participants affected / at risk) | 5/57 | 3/59
Other Adverse Events (participants affected / at risk) | 48/57 | 51/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Memantine (N=57) | Arm II - Placebo (N=59)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 2 (7)
Liver Dysfunction / Failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Retinal Tear (Eye disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Memantine (N=57) | Arm II - Placebo (N=59)
Back Pain (Musculoskeletal and connective tissue disorders) | 14 (54) | 12 (38)
Confusion (Psychiatric disorders) | 10 (21) | 5 (9)
Constipation (Gastrointestinal disorders) | 15 (31) | 13 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (69) | 27 (72)
Diarrhea (Gastrointestinal disorders) | 6 (12) | 10 (15)
Dizziness (Ear and labyrinth disorders) | 16 (25) | 10 (22)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (55) | 16 (40)
Fatigue (General disorders) | 33 (83) | 25 (66)
Headache (General disorders) | 19 (33) | 19 (33)
Hypertension (Cardiac disorders) | 13 (31) | 13 (37)
Renal and Urinary Disorder - Other (Renal and urinary disorders) | 1 (1) | 5 (15)
Somnolence (General disorders) | 13 (23) | 8 (17)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes